CLINICAL TRIAL: NCT04294953
Title: Efficacy of Perioperative Duloxetine as a Part of Multimodal Analgesia in Laparoscopic Colorectal Cancer Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mirna Ismail, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Duloxetine
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (I) (D) : (Duloxetine group) (Active Comparator)
  Interventions: Drug: Duloxetine
- Group (II) (P): (placebo group) (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Duloxetine — Each Patient will receive oral Duloxetine capsule 60mg at the night before operation(12hrs before surgery), the 2nd dose 60 mg Duloxetine capsule 1hr before operation and 3rd dose 60mg capsule after 24hrs postoperative
  Arms: Group (I) (D) : (Duloxetine group)
Drug: Placebo oral tablet — Each patient will receive a similar looking placebo capsule in the same time schedule. The placebo capsule will be prepared by hospital pharmacy to insure that active Duloxetine capsules will be indistinguishable from the placebo capsules contained starch
  Arms: Group (II) (P): (placebo group)

SUMMARY:
Our aim will be to evaluate the efficacy of perioperative Duloxetine in decreasing acute postoperative pain after laparoscopic colorectal cancer surgery and its role in reducing postoperative morphine requirements

DETAILED DESCRIPTION:
Abdominal surgery is usually associated with severe; wide spread post-operative pain. The greater propensity for pain and opioid-related side effects are likely contributing factors for poor postsurgical recovery, and it often results in significant pain and slow recovery. Although Opioids are considered the analgesics of choice to treat moderate to severe pain, their use carries the risk of side effects and hyperalgesia. Multimodal analgesia is advocated for perioperative pain management to reduce opioid use and its associated adverse effects. Multimodal analgesia can be achieved by combining different analgesics and different methods of administration, to provide better analgesia synergistically compared with conventional analgesia.Therefore, lower doses for each drug can be provided with fewer overall side-effects obtained from individual compounds.Serotonin and norepinephrine are involved in the modulation of endogenous analgesic mechanisms via descending inhibitory pain pathways in the brain and spinal cord. An increase in serotonin and norepinephrine may increase inhibition of nociceptive input and improve pain relief.

Duloxetine is a serotonin-norepinephrine reuptake inhibitor commonly prescribed for the treatment of major depression and anxiety. Duloxetine also has been used in the treatment of chronic pain conditions. There several reasons why duloxetine might improve postsurgical quality of recovery. First, systemic Duloxetine seems to have perioperative analgesic effects. In addition, as a serotonin-norepinephrine reuptake inhibitor, it is possible that the drug may prevent transient emotional problems that are common during the perioperative period. Lastly, the combination of less pain and better emotional status can result in better physical independence scores after surgery.

The main objective of the current study is to examine the effect of perioperative Duloxetine on postoperative pain after laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* aged 18-65 years and scheduled for laparoscopic colorectal surgery for cancer colon

Exclusion Criteria:

* unable to express their pain or patient refusal.
* allergy to the study drug
* an abnormal liver or renal function tests
* a chronic opioid abuser(> 3 mo), being on chronic gabapentin or pregabalin(> 3 mo)
* antidepressant drugs, patients with psychiatric disorders
* Pregnant females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 48 hours postoperative
  total morphine consumption(mg) in 48 hours if VAS score( Visual Analog Scale ) more than 3. score from 0 to 10 where 0 = no pain and 10 = the worst pain imaginable

SECONDARY OUTCOMES:
pain scores | 48 hours postoperative
  - pain scores ( theVAS score ).evaluation the pain using VAS ( Visual Analog Scale ) scored from 0 to 10 where 0 = no pain and 10 = the worst pain imaginable
first request of analgesia | 48 hours postoperative
  - the time of first request of analgesia (morphine) requirement postoperative
Postoperative sedation | 48 hours postoperative
  Postoperative sedation will be assessed using a modified observers. Assessment of alterness /sedation scale where 6= agitated to 0 = doesn't respond to deep stimulus.
Postoperative patient satisfaction | 48 hours postoperative
  Postoperative patient satisfaction will be measured using a numerical score of 1-4 (1= poor, 2= fair, 3= good, 4= very good) .

REFERENCES:
- [Background] Govil N, Parag K, Arora P, Khandelwal H, Singh A; Ruchi. Perioperative duloxetine as part of a multimodal analgesia regime reduces postoperative pain in lumbar canal stenosis surgery: a randomized, triple blind, and placebo-controlled trial. Korean J Pain. 2020 Jan 1;33(1):40-47. doi: 10.3344/kjp.2020.33.1.40. PMID 31888316
- [Background] Ho KY, Tay W, Yeo MC, Liu H, Yeo SJ, Chia SL, Lo NN. Duloxetine reduces morphine requirements after knee replacement surgery. Br J Anaesth. 2010 Sep;105(3):371-6. doi: 10.1093/bja/aeq158. Epub 2010 Jun 23. PMID 20573635
- [Background] Takmaz O, Bastu E, Ozbasli E, Gundogan S, Karabuk E, Kocyigit M, Dede S, Naki M, Kose F, Gungor M. Perioperative Duloxetine for Pain Management After Laparoscopic Hysterectomy: A Randomized Placebo-Controlled Trial. J Minim Invasive Gynecol. 2020 Mar-Apr;27(3):665-672. doi: 10.1016/j.jmig.2019.04.028. Epub 2019 Aug 30. PMID 31476481
- [Background] Attia JZ, Mansour HS. Perioperative Duloxetine and Etoricoxibto improve postoperative pain after lumbar Laminectomy: a randomized, double-blind, controlled study. BMC Anesthesiol. 2017 Dec 2;17(1):162. doi: 10.1186/s12871-017-0450-z. PMID 29197345